CLINICAL TRIAL: NCT03136133
Title: Effekt of Marine Peptide Supplementation on Recovery Following Endurance Cycling
Brief Title: Protein Supplements to Cyclists
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: Firmenich Bjørge Biomarine As (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/56
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Reconstitution After Bicycle Intervention

STUDY DESIGN:
Intervention Model Description: Crossover, placebo controlled
Who Masked: Participant
Masking Description: Protein drink With matching placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active protein drink (Active Comparator): Active protein drink
  Interventions: Dietary Supplement: Active protein drink
- Placebo drink (Placebo Comparator): Placebo drink
  Interventions: Dietary Supplement: Active protein drink

INTERVENTIONS:
Dietary Supplement: Active protein drink — Fish protein from cod to be used for man after Heavy excercise to restitute

SUMMARY:
To investigate the effect of marine peptide combined with dietary protein on the capacity to recover after exhaustive endurance cycling as measured by exercise capacity and blood glucose homeostasis.

DETAILED DESCRIPTION:
The current study uses cyclists as test subjects since they represent a physical demanding sport requiring both high endurance capacity and muscle strength. In the recovery phase following exhaustive physical activity there is a need both for rebuilding the muscle energy stores, for muscle repair and for compensatory muscle cell development. Therefore, marine peptide combined with dietary protein will be given in order to examine the capacity to recover after exhaustive endurance cycling.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed Consent
* The subject is a man between 40-50 years
* The subject has a body mass index (BMI) between 19-29
* Willing to comply with all study procedures and be available for the length of the study
* In good general health as judged by the physician at the screening visit

Exclusion Criteria:

* The subject has had surgery or trauma with significant blood loss or has donated blood within the last 3 months prior to the screening visit
* Diabetes type 1 or 2, or persistent high blood sugar levels
* The subject has tested positive for human immunodeficiency virus (HIV)
* Hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (anti-HCV)
* The subject has taken any investigational drugs within 1 month prior to screening
* Treated with antibiotics within 3 months prior to screening (oral, parenteral or rectal), but not spray or ointment
* Treated with steroids within 1 month prior to screening (including oral treatment)
* Treated with medication that effects the intestinal function such as, H2- protonpump inhibitors, diuretics, antiemetics, antidepressants, antacids,

Ages: 40 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-09-14 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in blood glucose compared to placebo | Change from baseline to every 30 minutes after dosing, for 2 hours

SECONDARY OUTCOMES:
Change in insulin-like peptide 5 compared to placebo | Change from baseline to every 30 minutes after dosing, for 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mjos I, Thorsen E, Hausken T, Lied E, Nilsen RM, Bronstad I, Edvardsen E, Frisk B. The effect of low dose marine protein hydrolysates on short-term recovery after high intensity performance cycling: a double-blinded crossover study. J Int Soc Sports Nutr. 2019 Oct 29;16(1):48. doi: 10.1186/s12970-019-0318-3. PMID 31665070